CLINICAL TRIAL: NCT06393998
Title: CO2 Supplement for Prophylaxis and Treatment of Acute Mountain Sickness Using Novel Device
Brief Title: CO2 Supplement for Treatment of Acute Mountain Sickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Key Laboratory of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Yuan-Ming Luo, Professor, State Key Laboratory of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020 037
Record Dates: First submitted 2024-04-20; First posted 2024-05-01 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Acute Mountain Sickness; High Altitude; Inhalation; Gas
Keywords: Acute mountain sickness; CO2 inhalation; central sleep apnea
MeSH Terms: conditions — Altitude Sickness; Respiratory Aspiration; Mucopolysaccharidosis IV; Sleep Apnea, Central

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing with CO2 during daytime and night at high altitude (Active Comparator): Subjects will sleep and perform exercise tests under inhalation of low concentration of CO2 supplied by a novel device at high altitude.
  Interventions: Device: Breathing with CO2 during daytime and night at high altitude
- Breathing with air during daytime and night at high altitude (Placebo Comparator): Subjects will sleep and perform exercise tests under inhalation of air at high altitude.
  Interventions: Device: Sleep and doing exercise test under inhalation of air

INTERVENTIONS:
Device: Breathing with CO2 during daytime and night at high altitude — Subjects wear the mask connecting to low dose CO2 supplied by a novel device during daytime and sleep dependent on the randomization once arriving high altitude.
  Other Names: Sleep and doing exercise test under inhalation of CO2
  Arms: Breathing with CO2 during daytime and night at high altitude
Device: Sleep and doing exercise test under inhalation of air — Subjects wear the mask connecting to air supplied by the novel device during daytime and sleep dependent on the randomization once arriving high altitude.
  Arms: Breathing with air during daytime and night at high altitude

SUMMARY:
It was reported that up to 76% people who rapidly ascend to the altitude higher than 4500 m without sufficient acclimatization will have AMS which often develops 6-8 hours after reaching at high altitude. AMS could be improved if there is no continuous ascent although central sleep apnea may persist much longer. It has also been well documented that exercise capacity was impaired at high altitude. Oxygen inhalation is the most effective treatment method, but it is impractical for outdoor activities because of the large volume required. There are some drugs such as acetazolamide, and ibuprofen for relieving AMS but side effects and inconsistent treatment effect made them to be difficulty for routine use. It is noted that adding CO2 might be useful for improvement of hypoxia and exercise ability and eliminating CSA. There is no available device which can accurately supply constant CO2 and is functionally free of dead space. We innovated a portable device with a special mask for supplement of CO2 for prophylaxis and treatment of AMS.

DETAILED DESCRIPTION:
Objective: To determine whether, after rapid ascent to high altitude the device could reduce the incidence and severity of AMS as defined by AMS scores, improve sleep quality and reduce central sleep apnea events.

Methods: A randomized placebo-controlled study will be performed in 36 healthy adults with no history of travelling to high altitude (>1000m) a year before the study. Subjects will be randomly and blindly given either CO2 mixed with air or air alone during daytime and sleep. Blood gases will be measured 30 minutes after inhalation of air or CO2. SaO2, heart rate, and respiratory rate will be recorded every two hours. AMS (Lake Louise Acute Mountain Sickness Score) will be recorded before and after sleep. PSG including diaphragm EMG would be recorded under CO2 or air. Exercise time, ventilation heart rate, respiratory rate, and SaO2 will be recorded and maximal load and peak ventilation will be measured during incremental cycle exercise with inhalation of CO2 or ambient air.

ELIGIBILITY:
Inclusion Criteria:

1. BMI less than 25kg/m2
2. normal lung function.
3. Healthy lowlanders (<500m) who have no history to travel to high altitude (>1000m) a year before the study.

Exclusion Criteria:

1. insomnia,
2. moderate or severe OSA based on PSG at sea level (AHI> 15 events/hr).
3. visited to an altitude >2500 m in the preceding year.
4. Currently using medicines for diabetes, hypertension et al.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-09-02 (Actual)

PRIMARY OUTCOMES:
Incidence rate of acute mountain sickness (AMS) | 72 hours
  Incidence rate of AMS based on Louis's scores under inhalation of CO2 and ambient air. The maximum score is 12 points, and a score greater than 3 indicates the presence of AMS.
The severity of AMS | 72 hours
  The severity of AMS based on Louis's scores under inhalation of CO2 and ambient air. A score of 3-5 indicates mild AMS, a score of 6-9 indicates moderate AMS and a score of 10-12 indicates severe AMS.

SECONDARY OUTCOMES:
Central sleep apnea index based on PSG | 72 hours
  Changes of central sleep apnea index under inhalation of CO2 and ambient air.
Sleep quality based on PSG | 72 hours
  Changes of sleep quality under inhalation of CO2 and ambient air.
Workload in the incremental ergometer test | 72 hours
  Changes of workload in the incremental ergometer test under inhalation of CO2 and ambient air.
Exercise duration in the incremental ergometer test | 72 hours
  Changes of exercise duration in the incremental ergometer test under inhalation of CO2 and ambient air.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanming Luo, PhD, Principal Investigator — Guangzhou Medical University
Locations (1):
- Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared after the paper of this study publishing.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be shared after the paper of this study publishing.
Access Criteria: After the paper of this study publishing